CLINICAL TRIAL: NCT07068568
Title: Dose Modulation Strategy of Sonidegib for Eye-Sparing Treatment of Locally Advanced Periocular Basal Cell Carcinoma
Brief Title: Dose-Modulated Sonidegib Therapy for Periocular Basal Cell Carcinoma
Acronym: BCC-Sonidegib
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Diego Strianese, Prof, Federico II University
Other Study IDs: AOU Federico II n. 2025/040325
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Basal Cell Cancer; Eyelid Tumor; Basal Cell Carcinoma (BCC); Basal Cell Carcinoma of the Head and Neck
Keywords: eyelid basal cell carcinoma; sonidegib
MeSH Terms: conditions — Neoplasms, Basal Cell; Eyelid Neoplasms; Carcinoma, Basal Cell | interventions — sonidegib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sonidegib-Treated laBCC Patients: This cohort includes adult patients diagnosed with locally advanced periocular basal cell carcinoma (laBCC) who were treated with oral Sonidegib (200 mg daily) at the University of Naples Federico II. All patients were considered unsuitable for surgical excision or radiotherapy due to the location or extent of the tumor, where standard approaches posed risks of vision loss or disfigurement. A personalized dose modulation strategy was applied based on treatment tolerance and clinical response, including temporary discontinuation or adjustment of dosing frequency. Patients were followed with regular dermatologic and ophthalmologic assessments to evaluate tumor response, functional outcomes, adverse events, and recurrence rates. The cohort reflects real-world clinical practice in managing complex periocular laBCC.
  Interventions: Drug: Sonidegib

INTERVENTIONS:
Drug: Sonidegib — Sonidegib was administered orally at a dose of 200 mg once daily as per approved guidelines. The intervention was applied in a real-world clinical setting to patients with histologically confirmed, locally advanced periocular basal cell carcinoma (laBCC) deemed unsuitable for surgical resection or radiotherapy due to the tumor's extent or proximity to critical ocular structures. A flexible, individualized dose modulation strategy was implemented to manage adverse effects and optimize patient adherence. Modifications included temporary treatment interruptions or reduced dosing frequency, tailored to each patient's clinical status and tolerance. The goal of the intervention was to achieve local tumor control while preserving ocular structures, visual function, and cosmetic appearance. All patients received regular multidisciplinary follow-up, including ophthalmologic and dermatologic assessments.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and clinical outcomes of a dose-modulation strategy of Sonidegib in adult patients with locally advanced periocular basal cell carcinoma (laBCC) who are not candidates for surgery or radiotherapy. The main questions it aims to answer are:

* Can dose-adjusted Sonidegib treatment preserve ocular function and avoid disfiguring surgery in laBCC patients?
* What is the rate of tumor response, recurrence, and adverse events during dose-modulated treatment?

Researchers will compare different dosing regimens based on treatment response, tolerability, and toxicity profiles to assess whether intermittent dosing or dose reductions can maintain clinical benefits while minimizing adverse effects.

This monocentric retrospective observational real-world evidence (RWE) study included 12 patients (8 male, 4 female; aged between 67 and 92 years; mean 83.25 years) with histologically confirmed periocular laBCC (staged T3-T4b) treated with sonidegib between 2021-2023 at the Oculoplasty Unit of the University of Naples Federico II. Eligible patients were those for whom conventional surgery or radiotherapy would result in loss of vision or unacceptable cosmetic outcomes.

Participants:

* Took Sonidegib orally, starting at 200 mg daily, with possible dose interruptions or reductions based on individual tolerance and tumor response.
* Underwent clinical and ophthalmologic evaluations every 4-6 weeks.
* Had imaging and dermatologic assessments to monitor tumor regression.
* Completed follow-up visits after treatment completion to assess long-term control and safety.

The results of this study aim to support an eye-sparing, patient-centered approach for complex periocular tumors.

DETAILED DESCRIPTION:
This monocentric, open-label, real-world study investigated the clinical efficacy and tolerability of Sonidegib, a selective Hedgehog pathway inhibitor, in the treatment of locally advanced periocular basal cell carcinoma (laBCC). The study specifically focused on patients for whom standard surgical or radiotherapy options were contraindicated due to the risk of vision loss, functional impairment, or unacceptable cosmetic outcomes.

A total of 12 adult patients with histologically confirmed periocular laBCC were enrolled at the Oculoplasty Unit of the University of Naples Federico II. Inclusion criteria targeted individuals with tumors in functionally or aesthetically sensitive locations-such as the eyelid margins, medial/lateral canthi, or deep orbital tissues-where conventional excision would require extensive, disfiguring surgery. All patients received oral Sonidegib 200 mg daily as first-line systemic therapy.

A dose-modulation strategy was implemented in response to adverse effects or individual tolerance, allowing temporary drug interruption or reduced-frequency administration. This personalized therapeutic approach aimed to preserve treatment adherence and quality of life while maintaining tumor control.

Patients were monitored through multidisciplinary follow-up visits at regular intervals, including dermatologic evaluation, photographic tumor documentation, and ophthalmologic assessments such as best-corrected visual acuity (BCVA), slit-lamp biomicroscopy, and fundus examination. Tumor response was assessed using clinical measurements and standardized criteria adapted for periocular anatomy.

The primary endpoint was the proportion of patients achieving disease control (complete response, partial response, or stable disease) without requiring exenteration or vision-threatening surgery. Secondary endpoints included time to response, duration of therapy, adverse event frequency and severity (graded per CTCAE), patient-reported functional and cosmetic outcomes, and post-treatment recurrence rates.

This study offers preliminary real-world evidence that Sonidegib, when administered with a flexible dosing strategy, can achieve significant therapeutic responses while minimizing toxicity in patients with complex periocular laBCC. The results support its role as an eye-sparing, function-preserving alternative to surgery in selected cases.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with histologically confirmed, locally advanced periocular basal cell carcinoma (laBCC)
* Tumor location or extent deemed unsuitable for surgical resection or radiotherapy due to high risk of orbital invasion, vision loss, or cosmetic disfigurement
* ECOG performance status 0-2
* Life expectancy ≥12 months
* Willing and able to comply with study procedures and follow-up assessments
* Provided written informed consent

Exclusion Criteria:

* Evidence of metastatic basal cell carcinoma
* Prior treatment with Hedgehog pathway inhibitors
* History of other malignancies within 5 years (except adequately treated non-melanoma skin cancer or carcinoma in situ)
* Severe hepatic or renal impairment
* Active systemic infection or uncontrolled medical conditions
* Pregnant or breastfeeding women
* Inability to undergo dermatologic or ophthalmologic evaluation due to physical or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of 12 adult patients with histologically confirmed, locally advanced periocular basal cell carcinoma (laBCC), all enrolled and treated at the Oculoplasty Unit of the University of Naples Federico II. All participants were treatment-naïve and presented with tumors unsuitable for surgical excision or radiotherapy due to the high risk of vision loss or anatomical disruption. The cohort included 8 males and 4 females, aged between 67 and 92 years, with a mean age of 83.25 years. The study was conducted in a real-world clinical setting and aimed to preserve ocular function and periocular anatomy through targeted oral therapy with Sonidegib.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Tumor Control Rate | From baseline to end of follow-up (ranging from 12 to 33 months)
  The primary outcome is the proportion of patients who achieved disease control, defined as complete response, partial response, or stable disease without requiring disfiguring surgery or orbital exenteration. Tumor response was assessed clinically and photographically during dermatologic evaluations, in combination with ophthalmologic monitoring for visual function preservation. Classification was based on established dermatologic and ophthalmologic criteria adapted to periocular anatomy. Treatment tolerability and the need for dose modulation were also recorded as part of the outcome analysis.

SECONDARY OUTCOMES:
Preservation of Visual Function and Ocular Structure | From treatment initiation through the final follow-up visit (12 to 33 months)
  This secondary outcome measures the proportion of patients maintaining functional vision and anatomical integrity of the eye during and after Sonidegib treatment. Evaluations included best-corrected visual acuity (BCVA), intraocular pressure, and slit-lamp and fundus examinations performed at baseline and at follow-up visits. Structural preservation was defined as avoidance of orbital invasion, enucleation, or significant deformation of periocular tissues. Changes in ocular function were documented and graded by the ophthalmology team to assess any Sonidegib-related ocular toxicity or surgery-preventing benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Strianese, MD, PhD, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Naples, Campania, Italy